CLINICAL TRIAL: NCT01564316
Title: Proteomics Study by Serum and Platelet With Neurodegeneration Disease Patients
Status: Terminated | Type: Observational
Why Stopped: The study has been terminated due to difficulties in gathering the patient samples.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-0505-148-016
Record Dates: First submitted 2012-03-11; First posted 2012-03-27 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Biomarker With Neurodegeneration Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum:10ml
  WHO: neurodegeneration patients and control group include dementia patients visited the part of neurology.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- neurodegeneration patients: •neurodegeneration patients and control group include dementia patients visited the part of neurology

SUMMARY:
Using to method of Proteomics, for aims to conquer intractable disease, try to access variety experiment. Biomarker is necessary to develop new diagnosis method and target of treatment.

DETAILED DESCRIPTION:
Following Seoul National University Hospital Institutional Review Board approval, obtain serum and platelet with neurodegeneration patients and control group visited the part of neurology, there'll be analysis to differentiate each other diseases use to method Proteomics. Biomarker will be screening via 1D/2D analysis, Mass analysis, database searching- the MASCOT search tool, SWISS-PROT and etc.

ELIGIBILITY:
Inclusion Criteria:

* neurodegeneration patients and control group include dementia patients visited the part of neurology.
* over the age of 18
* when participants can understand subject of this study
* Total point of Mini Mental state exam(MMSE)should be Under 26 include MCI (mild cognitive impairment) and over GDS score 3points.

exclusion criteria:

* under eighteen years of age
* when participants cannot understand subject of this study
* cannot accept this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: neurodegeneration patients group include dementia patients visited the part of neurology.
  (almost after diagnosis)
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2005-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manho Kim, Professor, Study Director — Seoul National University Hospital
Locations (1):
- Department of Neurology, Seoul National University Hospital, Seoul, Seoul, South Korea